CLINICAL TRIAL: NCT05606900
Title: Eye Movements Desensitization and Reprocessing (EMDR) Intervention in Preventing Craving in Alcohol Use Disorder: Randomized Controlled Study
Brief Title: Eye Movements Desensitization and Reprocessing Intervention in Preventing Craving in Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Yagmur Callak, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-8.2
Record Dates: First submitted 2022-10-30; First posted 2022-11-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder; Alcohol Craving
Keywords: alcohol use disorder; alcohol craving; eye movement desensitization reprocessing; emdr; controlled trial
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: This study was designed as an open-label randomized controlled trial.
Who Masked: Investigator
Masking Description: The randomisation of patients to one of the study arms will be carried out by another researcher other than the researcher who will practice the intervention. With this masking method, it is planned to assign the patients to the groups without any bias of the psychotherapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment group (Experimental): Twenty volunteer patients between the ages of 18-65 who applied to the addiction polyclinic and were diagnosed with alcohol use disorder (AUD) constitute the sample of the experimental group. In addition to the standard alcohol addiction treatment (TAU) applied in the addiction polyclinic, the patients in the experimental group will be given addiction-focused eye movements, desensitization and reprocessing (AF-EMDR) psychotherapy. AF-EMDR consists of 3 sessions, with a total duration of 3 weeks. Each session will last between 1 and 1 and a half hours, depending on individual differences. Psychotherapy sessions will be conducted as face-to-face and individual sessions. TAU includes the medical treatment for AUD and motivational interviews if necessary, administered by the psychiatrist in the addiction polyclinic, where the research is conducted. Structured psychotherapy is not used in TAU practice.
  Interventions: Behavioral: addiction-focused eye movements desensitization and reprocessing (AF-EMDR)
- Control group (No Intervention): The sample of the control group consists of 20 volunteer patients between the ages of 18-65 who applied to the addiction polyclinic and were diagnosed with alcohol use disorder (AUD). Patients in the control group will be given standard treatment of alcohol use disorder (TAU). The duration and dosage of TAU are regulated by the psychiatrist in the polyclinic specific to the patient. During the duration of AF-EMDR to the experimental group, patients in the control group will be on the waiting list and will not receive AF-EMDR intervention. If AF-EMDR intervention is concluded as beneficial for the patients in the experimental group after the analysis of the final measurements (1-month follow-up measurements), the same AF-EMDR intervention will be applied to the patients in the control group.

INTERVENTIONS:
Behavioral: addiction-focused eye movements desensitization and reprocessing (AF-EMDR) — AF-EMDR includes desensitization and functional reprocessing of the targeted memory or the moment with lateral eye movements. In each session of the psychotherapy, which will be applied as 3 sessions, a memory or a moment that causes alcohol craving will be practised. The processing will continue until the patient becomes desensitized to the memory or the moment that cause the craving. In the first session, a memory of craving will be discussed, in the second session a current trigger that causes craving, and in the third session, a moment that is thought to cause craving in the future will be focused.
  Arms: Experiment group

SUMMARY:
This study is conducted to examine the effect of a psychotherapy model that is expected to affect alcohol cravings in adults aged 18-65 years who are being treated for alcohol use disorder at a clinic. The psychotherapy intervention is expected to affect other variables such as clinical symptom level, self-efficacy level, and functionality level. This protocol is called addiction-focused eye movement desensitization and reprocessing (addiction-focused EMDR). Patients found suitable for the study will be divided into experimental and control groups. The intervention will be applied to the experimental group and not to the control group. At the end of the intervention, the effect of the intervention primarily on the level of craving will be compared with that of the control group. The intervention is expected to reduce the level of craving. The intervention is expected to have an impact on the other variables mentioned as well.

DETAILED DESCRIPTION:
The main purpose of this study is to examine the change in craving frequency, craving severity, and level of control over craving in adults who applied to an addiction clinic and diagnosed with alcohol use disorder after having the intervention of addiction-focused eye movements and desensitization and reprocessing (addiction-focused EMDR) therapy. The sub-objectives of the study are to monitor the changes in the clinical symptoms, self-efficacy and general functionality levels of addicted individuals receiving addiction-focused EMDR therapy. The research will be carried out at Ege University Substance Abuse, Toxicology and Pharmaceutical Sciences Institute Addiction Polyclinic. The population of the research consists of individuals between the ages of 18-65 who applied to Ege University Substance Abuse, Toxicology and Pharmaceutical Sciences Institute Addiction Polyclinic and were diagnosed with alcohol use disorder. In order to estimate the effect size and sample size of the research, the data obtained from a reference research were used due to its suitability for the design, purpose and primary output of the research, and the calculations were made on G Power 3.1. Confidence interval was taken as 95% (p<0.05) and power was determined as 80%. As a result of the calculation, the effect size was found to be f: 0.42 and the total number of samples was determined as 30. According to the previous research, the sample loss rate was reported as 33%. When the estimated sample loss at a similar rate is added to the research, the final sample number was determined as 40 patients, 20 patients in the control group and 20 patients in the intervention group. Sociodemographic Form created by the researcher to obtain information about the patients' age, gender, past diagnosis, treatment histories, and medical diseases; Alcohol Use Disorders Identification Test to measure the risk level of alcohol use; Penn Alcohol Craving Scale to measure craving severity and frequency; Craving Experience Scale to measure the level of control over craving; Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) Self-Rated Level 1 Cross-Cutting Symptom Scale to measure the level of clinical symptoms; Childhood Trauma Questionnaire; General Self-Efficacy Scale; The General Assessment of Functioning Scale to measure the level of functionality in the social, occupational and psychological domains will be used to gather the data. Statistical analysis of the data will be performed in Statistical Package for the Social Sciences (SPSS). Repeated measures analysis of variance (ANOVA) test will be used to calculate whether there is a difference between the experimental and control groups in terms of measured variables. The significance value (p) will be taken as 0.05. The results will be presented in tables, reported and discussed within the light of the literature.

Research Duration

The total duration of the research is planned to be 15 months between October 2022 and December 2023. The stages of the research were planned according to weeks (W). The stages of the research and the plan according to the weeks are as follows:

1. Sample screening (October 2022, W1-W4) 2. Evaluation session and pre-measurements (October 2022, W2-W4) 3. Randomization and research groups (November 2022, W5-W6) 4. Informing the participants (November 2022, W5-W6) 5. Intervention (psychotherapy sessions) (November 2022-December 2022, W7-W12) 6. Post-measurements (December 2022-January 2023, W11-W13) 7. Follow-up measurements (January 2023-February 2023, W15-W17) 8. Analyzing the data (February 2023, W18-W20) 9. Intervention in the control group (March 2023-April 2023, W22-W29) 10. Reporting (May 2023-December 2023, W30-W60)

1. Sample Screening Face-to-face or telephone interviews will be conducted with patients who have applied to Ege University Substance Abuse, Toxicology and Pharmaceutical Sciences Institute Addiction Polyclinic and diagnosed with alcohol use disorder. Meeting appointment for a face-to-face evaluation will be made with the patients who are interested in the research. Preliminary interviews will continue and appointments will be made until the sufficient number of samples is reached. Sample screening and interviews with volunteer patients are expected to be conducted and completed between the first and fourth weeks of October 2022.
2. Evaluation Session and Pre-measurements The steps in the evaluation session (clinical evaluation) can be listed as follows.

   Patients who participate in the evaluation interview will be informed in detail about the content of the research. It will be stated that the participants will be randomly divided into two groups via a randomisation program by another researcher. Patients who accept to participate in the research will have to sign a standard informed consent form and a copy of which will be given to them.

   The anamnesis of the patients who voluntarily agreed to participate in the research will be taken. Anamnesis information will be recorded in the Sociodemographic Form prepared by the primary researcher.

   All scales (Alcohol Use Disorders Identification Test, Penn Alcohol Craving Scale, Craving Experience Scale, DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Scale, Childhood Trauma Questionnaire, General Self-Efficacy Scale, The General Assessment of Functioning Scale) will be applied to the patients in company with the primary researcher. These measurements are the pre-measurements of the research (t0).

   Patients will be informed to be contacted again in order to inform them about which group they are in, before the session will be ended.
3. Randomization and Research Groups After the evaluation session, patients who meet the criteria for inclusion in the research will be determined according to the information obtained from the measurement tools. Each participant will be assigned a protocol number. Participants will be assigned to one of the experimental and control groups by stratified randomization method over protocol numbers. Stratified randomization assignments will be based on homogeneity of age, gender, severity of addiction, severity of craving, past treatment history, severity of clinical symptoms, and severity of childhood trauma. Randomization process will be performed by another researcher other than the primary researcher who will perform the intervention so blindness will be ensured in the randomization of the research groups. If sufficient sample size (N=40) is not reached at the initial interviews, randomizations will be made in groups. Depending on the intensity and duration of reaching the participants, 4 groups of 10 participants each, 2 groups of 20 participants each, or 4 groups of 10 participants each will be randomized separately.
4. Informing the Participants After the patients are divided into research groups, first psychotherapy session will be scheduled by communicating with the participants in the experimental group. Participants in the control group will be contacted and informed that they are on the waiting list. Patients who are determined to be unsuitable for participation in the research in accordance with the exclusion criteria will be contacted and informed that they will not be able to participate in the research.
5. Intervention (Psychotherapy Sessions): Addiction-Focused Eye Movement Desensitization Reprocessing Psychotherapy (AF-EMDR) The AF-EMDR intervention will be carried out in accordance with the standard protocol, with an average of 1 week interval between each psychotherapy session, on the dates and times determined with the patients in the experimental group. Session duration is between 60-90 minutes. The intervention, which will consist of a total of three sessions, is planned to end within a period of 3 weeks, unless otherwise occurs (such as the participant's postponing the session).

   Each psychotherapy session will be based on addiction-focused processing of the standard EMDR protocol. In the first session a memory of alcohol craving, in the second session a current trigger for craving, and in the last session a future craving situation will be processed. The content to be processed in sessions will be determined according to the information received from the patients.

   Participants who attend only one or two psychotherapy sessions will not be deemed to have completed the intervention. Participants who attend all three sessions will be deemed to have completed the intervention.

   Standard treatment (TAU): During the period of AF-EMDR intervention, all patients in the experimental and control groups will continue to receive TAU from the addiction outpatient clinic. The content and duration of TAU will be determined for each patient by the clinic's psychiatrist. TAU basically consists of medical treatment and motivational interviews when necessary.
6. Post-measurements and Follow-up Measurements DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Scale, Penn Alcohol Craving Scale, Craving Experience Scale, General Self-Efficacy Scale and General Assessment of Functioning will be used as measurement tools for post-measurements and follow-up measurements. Measurements will be made simultaneously for all patients in the experimental and control groups.

   1. Post-measurements (t1) will be made 4 weeks after the start of the interventions (the date of the first psychotherapy session will be considered as the intervention start date).
   2. Follow-up-measurements (t2) will be made 4 weeks after the post-measurements.
7. Analyzing the Data After the follow-up measurements are completed, the data obtained with the data collection tools will be analyzed. Experimental and control groups will be compared in terms of dependent variables of the research.
8. Intervention in the Control Group As a result of the analysis, if the participants in the experimental group benefit from the AF-EMDR intervention, the same intervention will be applied to the participants in the control group for ethical reasons.
9. Reporting The research process and the findings will be reported and presented in tables. The reporting part is the final stage of the research.

ELIGIBILITY:
Inclusion Criteria:

* Having the criteria for the diagnosis of alcohol use disorder according to DSM-5,
* Continuing or completing the standard treatment applied in the addiction clinic,
* Being between the ages of 18-65.

Exclusion Criteria:

* As a result of the clinical interview, meeting the criteria for any of the disorders included in the classifications of:

  1. "Bipolar and related disorders" with psychotic features,
  2. "Depression disorders" with psychotic features,
  3. "Dissociative disorders" such as depersonalization, derealization, dissociative identity disorder,
  4. "Schizophrenia spectrum and disorders leading to psychosis" such as schizophrenia, schizotypal personality disorder, schizoaffective disorder,
* Receiving any psychological or medical treatment other than the standard alcohol use disorder treatment administered in the Addiction Polyclinic,
* Having at least one of cardiovascular diseases, vertigo, epilepsy or eye diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of alcohol craving assessed by Penn Alcohol Craving Scale | The change scores of the frequency of alcohol craving between the control and the experiment groups will be compared between the baseline measure (t0) and the intervention completion (t1)(estimated to be 8 weeks).
  This outcome refers to the change in scores of the frequency of alcohol craving obtained from measurements at two time points between experiment and control groups. Penn Alcohol Craving Scale is the measurement tool to measure the craving frequency.
Frequency of alcohol craving assessed by Penn Alcohol Craving Scale | The change scores of the frequency of alcohol craving between the control and the experiment groups will be compared between the intervention completion (t1)(estimated to be 8 weeks) and 4-week follow-up (t2).
  This outcome refers to the change in scores of the frequency of alcohol craving obtained from measurements at two time points between experiment and control groups. Penn Alcohol Craving Scale is the measurement tool to measure the craving frequency.
Severity of alcohol craving assessed by Penn Alcohol Craving Scale | The change scores of the severity level of alcohol craving between the control and the experiment groups will be compared between the baseline measure (t0) and the intervention completion (t1)(estimated to be 8 weeks).
  This outcome refers to the change in scores of the severity level of alcohol craving obtained from measurements at two time points between experiment and control groups. Penn Alcohol Craving Scale is the measurement tool to measure the level of craving severity.
Severity of alcohol craving assessed by Penn Alcohol Craving Scale | The change scores of the severity level of alcohol craving between the control and the experiment groups will be compared between the intervention completion (t1)(estimated to be 8 weeks) and 4-week follow-up (t2).
  This outcome refers to the change in scores of the severity level of alcohol craving obtained from measurements at two time points between experiment and control groups. Penn Alcohol Craving Scale is the measurement tool to measure the level of craving severity.
Control level over alcohol craving assessed by Craving Experience Scale | The change scores of the control level over alcohol craving between the control and the experiment groups will be compared between the baseline measure (t0) and the intervention completion (t1)(estimated to be 8 weeks).
  This outcome refers to the change in scores of the control level over alcohol craving obtained from measurements at two time points between experiment and control groups. Craving Experience Scale is the measurement tool to measure the level of control over craving.
Control level over alcohol craving assessed by Craving Experience Scale | The change scores of the control level over alcohol craving between the control and the experiment groups will be compared between the intervention completion (t1)(estimated to be 8 weeks) and 4-week follow-up (t2).
  This outcome refers to the change in scores of the control level over alcohol craving obtained from measurements at two time points between experiment and control groups. Craving Experience Scale is the measurement tool to measure the level of control over craving.

SECONDARY OUTCOMES:
Clinical symptom levels assessed by Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) Self-Rated Level 1 Cross-Cutting Symptom Scale | The change scores of the clinical symptoms between the control and the experiment groups will be compared between the baseline measure (t0) and the intervention completion (t1)(estimated to be 8 weeks).
  This outcome refers to the difference in scores of the clinical symptoms including depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, and dissociation obtained from measurements at two time points between experiment and control groups. Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) Self-Rated Level 1 Cross-Cutting Symptom Scale is the measurement tool to measure the level of clinical symptoms. The total score in each sub-domain differs and yet 2 points and above in each sub-domain indicates moderate severity except the domains of suicidal ideation and psychosis of which 1 point is considered severe.
Clinical symptom levels assessed by Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) Self-Rated Level 1 Cross-Cutting Symptom Scale | The change scores of the clinical symptoms between the control and the experiment groups will be compared between the intervention completion (t1)(estimated to be 8 weeks) and 4-week follow-up (t2).
  This outcome refers to the difference in scores of the clinical symptoms including depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, and dissociation obtained from measurements at two time points between experiment and control groups. Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) Self-Rated Level 1 Cross-Cutting Symptom Scale is the measurement tool to measure the level of clinical symptoms. The total score in each sub-domain differs and yet 2 points and above in each sub-domain indicates moderate severity except the domains of suicidal ideation and psychosis of which 1 point is considered severe.
Self-efficacy level assessed by General Self-Efficacy Scale | The change scores of the level of self-efficacy between the control and the experiment groups will be compared between the baseline measure (t0) and the intervention completion (t1)(estimated to be 8 weeks).
  This outcome refers to the chance in scores of the self-efficacy obtained from measurements at two time points between experiment and control groups. General Self-Efficacy Scale is the measurement tool to measure the level of self-efficacy.
Self-efficacy level assessed by General Self-Efficacy Scale | The change scores of the level of self-efficacy between the control and the experiment groups will be compared between the intervention completion (t1)(estimated to be 8 weeks) and 4-week follow-up (t2).
  This outcome refers to the chance in scores of the self-efficacy obtained from measurements at two time points between experiment and control groups. General Self-Efficacy Scale is the measurement tool to measure the level of self-efficacy.
General functioning level assessed by The General Assessment of Functioning Scale | The change scores of the level of general functionality between the control and the experiment groups will be compared between the baseline measure (t0) and the intervention completion (t1)(estimated to be 8 weeks).
  This outcome refers to the change in scores of the general functionality in the social, occupational and psychological domains obtained from measurements at two time points between experiment and control groups. The General Assessment of Functioning Scale is the measurement tool to measure the level of general functioning.
General functioning level assessed by The General Assessment of Functioning Scale | The change scores of the level of general functionality between the control and the experiment groups will be compared between the intervention completion (t1)(estimated to be 8 weeks) and 4-week follow-up (t2).
  This outcome refers to the change in scores of the general functionality in the social, occupational and psychological domains obtained from measurements at two time points between experiment and control groups. The General Assessment of Functioning Scale is the measurement tool to measure the level of general functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Zeki Yuncu, Prof, Study Director — Ege University
Locations (1):
- Ege University, Substance Abuse, Toxicology and Pharmaceutical Sciences Institute, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boening JA. Neurobiology of an addiction memory. J Neural Transm (Vienna). 2001;108(6):755-65. doi: 10.1007/s007020170050. PMID 11478425
- [Background] Carletto S, Oliva F, Barnato M, Antonelli T, Cardia A, Mazzaferro P, Raho C, Ostacoli L, Fernandez I, Pagani M. EMDR as Add-On Treatment for Psychiatric and Traumatic Symptoms in Patients with Substance Use Disorder. Front Psychol. 2018 Jan 11;8:2333. doi: 10.3389/fpsyg.2017.02333. eCollection 2017. PMID 29375445
- [Background] Castelnuovo G, Fernandez I, Amann BL. Editorial: Present and Future of EMDR in Clinical Psychology and Psychotherapy. Front Psychol. 2019 Sep 27;10:2185. doi: 10.3389/fpsyg.2019.02185. eCollection 2019. No abstract available. PMID 31611832
- [Background] Hase M, Schallmayer S, Sack M. EMDR reprocessing of the addiction Memory: pretreatment, posttreatment, and 1-month follow-up. Journal of EMDR Practice and Research. 2008; 2(3):170-179. doi: 10.1891/1933-3196.2.3.170.
- [Background] Littel M, van den Hout MA, Engelhard IM. Desensitizing Addiction: Using Eye Movements to Reduce the Intensity of Substance-Related Mental Imagery and Craving. Front Psychiatry. 2016 Feb 8;7:14. doi: 10.3389/fpsyt.2016.00014. eCollection 2016. PMID 26903888
- [Background] Luber M. Eye Movement Desensitization and Reprocessing (EMDR) Scripted Protocols: Special Populations. New York: Springer Publishing Company. 2010.
- [Background] Markus W, Hornsveld HK, Burk WJ, de Weert-van Oene GH, Becker ES, DeJong CAJ. Addiction-Focused Eye Movement Desensitization and Reprocessing Therapy as an Adjunct to Regular Outpatient Treatment for Alcohol Use Disorder: Results From a Randomized Clinical Trial. Alcohol Clin Exp Res. 2020 Jan;44(1):272-283. doi: 10.1111/acer.14249. Epub 2019 Dec 17. PMID 31758556
- [Background] Markus W, de Weert-van Oene GH, Becker ES, DeJong CA. A multi-site randomized study to compare the effects of Eye Movement Desensitization and Reprocessing (EMDR) added to TAU versus TAU to reduce craving and drinking behavior in alcohol dependent outpatients: study protocol. BMC Psychiatry. 2015 Mar 18;15:51. doi: 10.1186/s12888-015-0431-z. PMID 25884223
- [Background] Perez-Dandieu B, Tapia G. Treating Trauma in Addiction with EMDR: A Pilot Study. J Psychoactive Drugs. 2014 Oct-Dec;46(4):303-9. doi: 10.1080/02791072.2014.921744. PMID 25188700
- [Background] Robbins TW, Ersche KD, Everitt BJ. Drug addiction and the memory systems of the brain. Ann N Y Acad Sci. 2008 Oct;1141:1-21. doi: 10.1196/annals.1441.020. PMID 18991949
- [Background] Shapiro F. The role of eye movement desensitization and reprocessing (EMDR) therapy in medicine: addressing the psychological and physical symptoms stemming from adverse life experiences. Perm J. 2014 Winter;18(1):71-7. doi: 10.7812/TPP/13-098. PMID 24626074
- [Background] Shapiro F. Eye Movement Desensitization and Reprocessing (EMDR) Therapy: Basic Principles, Protocols, and Procedures. New York: Guilford Publications. 2007.
- [Background] Sinha R. New findings on biological factors predicting addiction relapse vulnerability. Curr Psychiatry Rep. 2011 Oct;13(5):398-405. doi: 10.1007/s11920-011-0224-0. PMID 21792580
- See also: World Health Organization (2013). Guidelines for the management of conditions that are specifically related to stress. — http://apps.who.int/iris/bitstream/handle/10665/85119/9789241505406_eng.pdf;jsessionid$=$A87FC4134F1F50FE3F66C587868D2F32?sequence$=$1.
- See also: World Health Organization (2018). Global status report on alcohol and health. — http://apps.who.int/iris/bitstream/handle/10665/274603/9789241565639-eng.pdf?ua=1.